CLINICAL TRIAL: NCT02257177
Title: A Placebo-controlled RCT in HV's Investigating the Safety, Tolerability and PK (Pharmacokinetic) of TD139, a Galectin-3 Inhibitor, Followed by an Expansion Cohort Treating Subjects With Idiopathic Pulmonary Fibrosis (IPF)
Brief Title: RCT (Randomized Control Trial) of TD139 vs Placebo in HV's (Human Volunteers) and IPF Patients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Galecto Biotech AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GB-HV-01
Record Dates: First submitted 2014-09-29; First posted 2014-10-06 (Estimated); Results first posted 2021-04-08 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2021-03

CONDITIONS: Idiopathic Pulmonary Fibrosis
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (11):
- 0.15 mg TD139 (Part 1) (Active Comparator): 4 Healthy Subjects are administered a single dose of 0.15mg TD139 inhaled as a dry powder in a fasted state. Each cohort will include a dose leader volunteer to be dosed a day before the rest of the cohort, followed by the remaining 3 subjects who will be dosed approximately 24 hours later.
  Interventions: Drug: Inhaled TD139
- 1.5 mg TD139 (Part 1) (Active Comparator): 4 Healthy Subjects are administered a single dose of 1.5mg TD139 inhaled as a dry powder in a fasted state. Each cohort will include a dose leader volunteer to be dosed a day before the rest of the cohort, followed by the remaining 3 subjects who will be dosed approximately 24 hours later.
  Interventions: Drug: Inhaled TD139
- 3 mg TD139 (Part 1) (Active Comparator): 4 Healthy Subjects are administered a single dose of 3mg TD139 inhaled as a dry powder in a fasted state. Each cohort will include a dose leader volunteer to be dosed a day before the rest of the cohort, followed by the remaining 3 subjects who will be dosed approximately 24 hours later.
  Interventions: Drug: Inhaled TD139
- 10 mg TD139 Part 1 (Active Comparator): 4 Healthy Subjects are administered a single dose of 10mg TD139 inhaled as a dry powder in a fasted state. Each cohort will include a dose leader volunteer to be dosed a day before the rest of the cohort, followed by the remaining 3 subjects who will be dosed approximately 24 hours later.
  Interventions: Drug: Inhaled TD139
- 20 mg TD139 Part 1 (Active Comparator): 4 Healthy Subjects are administered a single dose of 20mg TD139 inhaled as a dry powder in a fasted state. Each cohort will include a dose leader volunteer to be dosed a day before the rest of the cohort, followed by the remaining 3 subjects who will be dosed approximately 24 hours later.
  Interventions: Drug: Inhaled TD139
- 50 mg TD139 Part 1 (Active Comparator): 4 Healthy Subjects are administered a single dose of 50mg TD139 inhaled as a dry powder in a fasted state. Each cohort will include a dose leader volunteer to be dosed a day before the rest of the cohort, followed by the remaining 3 subjects who will be dosed approximately 24 hours later.
  Interventions: Drug: Inhaled TD139
- Placebo Part 1 (Placebo Comparator): 12 Healthy Subjects are administered placebo inhaled as a dry powder in a fasted state. Each cohort will include a dose leader volunteer to be dosed a day before the rest of the cohort, followed by the remaining 3 subjects who will be dosed approximately 24 hours later.
  Interventions: Drug: Placebo
- 0.3 mg TD139 Part 2 (Active Comparator): 5 Patients with IPF are administered a single dose of 0.3mg TD139 once daily for 14 days inhaled as a dry powder.
  Interventions: Drug: Inhaled TD139
- 3 mg TD139 Part 2 (Active Comparator): 5 Patients with IPF are administered a single dose of 3mg TD139 once daily for 14 days inhaled as a dry powder.
  Interventions: Drug: Inhaled TD139
- 10 mg TD139 Part 2 (Active Comparator): 5 Patients with IPF are administered a single dose of 10mg TD139 once daily for 14 days inhaled as a dry powder.
  Interventions: Drug: Inhaled TD139
- Placebo Part 2 (Placebo Comparator): 9 Patients with IPF are administered placebo inhaled as a dry powder.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Inhaled TD139 — DPI Galectin-3 inhibitor
  Other Names: TD139
  Arms: 0.15 mg TD139 (Part 1); 0.3 mg TD139 Part 2; 1.5 mg TD139 (Part 1); 10 mg TD139 Part 1; 10 mg TD139 Part 2; 20 mg TD139 Part 1; 3 mg TD139 (Part 1); 3 mg TD139 Part 2; 50 mg TD139 Part 1
Drug: Placebo — DPI placebo
  Other Names: inhaled placebo
  Arms: Placebo Part 1; Placebo Part 2

SUMMARY:
This study will be divided into 2 parts. Part 1 is a randomized, double-blind, single centre, placebo-controlled, single ascending dose (SAD) phase I study designed to assess the safety, tolerability, PK and PD (Pharmacodynamic) of TD139 in up to 36 healthy male subjects. Part 2 will be a randomized, double-blind, multi-centre, placebo-controlled, multiple dose expansion cohort, designed to assess the safety, tolerability, PK and PD of TD139 in up to 24 male subjects and female subjects of non child-bearing potential with IPF.

DETAILED DESCRIPTION:
Up to 6 cohorts of 6 subjects will be randomly assigned in a blinded fashion to receive either a single dose of TD139 or matching placebo via DPI (dry powder inhaler) in an ascending dose fashion.

A single cohort of up to 24 patients will be randomly assigned in a blinded fashion to receive a single dose of TD139 or placebo via DPI once daily for 14 days in a 2:1 TD139 to placebo ratio. The dose of TD139 selected will be based on data from Part 1 and on pre-clinical efficacy and safety data.

ELIGIBILITY:
Part 1 Inclusion Criteria

* Healthy male subjects aged between 18 and 55 years of age.
* Male subject willing to use a condom, if applicable (unless anatomically sterile or where abstaining from sexual intercourse is in line with the preferred and usual lifestyle of the subject) from the Day 1 dose of study medication until 3 months afterwards.
* Subject with a body weight of at least 50 kg and a body mass index (BMI) within the range of 18 35 kg/m2. BMI = Body weight (kg) / [Height (m)]2.
* Subject with no clinically significant abnormal serum biochemistry, haematology and urine examination values within 28 days of the Day 1 dose of study medication.
* Subject with a negative urinary drugs of abuse screen, determined within 28 days of the Day 1 dose of study medication, (N.B. a positive alcohol result may be repeated at the discretion of the Investigator).
* Subject with negative human immunodeficiency virus (HIV) and hepatitis B surface antigen (Hep B) and hepatitis C virus antibody (Hep C) results.
* Subject with no clinically significant abnormalities in 12 lead ECG determined within 28 days of the Day 1 dose of study medication.
* Subjects were non smokers or former smokers (having ceased smoking for at least 6 months).
* Subjects with no clinically significant impairment in oxygen saturation.
* Subject satisfied a medical examiner about their fitness to participate in the study.
* Subject provided written informed consent to participate in the study.
* Subject was available to complete the study (including all follow up visits).

Confirmed at Baseline / Prior to First Dose:

* Subject continued to meet all screening inclusion criteria.
* Subject with a negative urinary drugs of abuse screen (including alcohol) prior to dosing.

Exclusion Criteria

* A clinically significant illness or surgery within 8 weeks prior to the Day 1 dose of study medication.
* Significant medical history that, in the Investigator's opinion, may have adversely affected participation.
* History of allergy or significant adverse reaction to drugs similar to the investigational drug, to nicotine, or to cholinergic drugs or to any drugs with a similar chemical structure.
* History of hypersensitivity (anaphylaxis, angioedema) to any drug.
* Use of any drug known to induce or inhibit hepatic drug metabolism, within 30 days prior to the Day 1 dose of study medication.
* Use of medications known to prolong QT/QTc interval within 14 days prior to the Day 1 dose of study medication.
* Any clinically significant findings of physical examination or laboratory findings at screening.
* A clinically significant history of drug or alcohol abuse.
* Receipt of regular/over the counter medication within 14 days of the Day 1 dose of study medication that may have had an impact on the safety and objectives of the study (at the Investigator's discretion).
* Evidence of renal, hepatic, central nervous system, respiratory, cardiovascular or metabolic dysfunction.
* Inability to communicate well with the Investigator (i.e., language problem, poor mental development or impaired cerebral function).
* Participation in a New Chemical Entity clinical study within the previous 4 months or a marketed drug clinical study within the previous 3 months. (N.B. washout period between studies is defined as the period of time elapsed between the last dose of the previous study and the first dose of the next study).
* Donation of 450 mL or more blood within the previous 3 months.

Confirmed at Baseline / Prior to First Dose:

* Development of any exclusion criteria since screening.
* Receipt of any medication since screening that may have had an impact on the safety and objectives of the study (at the Investigator's discretion).

Part 2 Inclusion Criteria

* Male patient or female patient of non childbearing potential with IPF.
* Male patient willing to use a condom, if applicable (unless anatomically sterile or where abstaining from sexual intercourse was in line with the preferred and usual lifestyle of the patient) from the first dose until at least 3 months after receiving the last dose of IMP.
* Aged between 45 and 85 years of age.
* With a forced vital capacity (FVC) ≥ 45% predicted and forced expiratory volume in 1 second (FEV1)/FVC ratio ≥ 0.7.
* Oxygen saturation > 90% by pulse oximetry while breathing ambient air at rest.
* Diffusing capacity of lungs for carbon monoxide (DLCO) > 25%.
* Had adequate organ function and a clinical diagnosis consistent with IPF prior to screening (based on the American Thoracic Society, the European Respiratory Society, the Japanese Respiratory Society and the Latin American Thoracic Association (ATS/ERS/JRS/ALAT) consensus criteria. The diagnosis would ordinarily have been confirmed at a multidisciplinary team meeting where the high resolution computed tomography (HRCT) findings in particular would have been discussed with a radiologist with respiratory expertise.
* Able to undergo BAL.
* Provided written informed consent to participate in the study.
* Available to complete the study (including all follow up visits).
* Negative urinary drugs of abuse screen, determined within 28 days of the first dose of IMP (N.B. a positive alcohol result could have been repeated at the discretion of the Investigator).
* Negative human immunodeficiency virus (HIV) and hepatitis B surface antigen (Hep B) and hepatitis C virus antibody (Hep C) results.
* No clinically significant abnormalities in 12 lead ECG determined within 28 days of the first dose of IMP.

Confirmed at Baseline / Prior to First Dose:

* Patient continued to meet all screening inclusion criteria. Exclusion Criteria
* Any condition that made the patient at unacceptable risk for bronchoscopy.
* Active cigarette smoking (defined as smoking more than 3 cigarettes daily within the last 6 months).
* Presence of a significant co morbidity felt to limit life expectancy to less than 12 months.
* HRCT pattern showing emphysema more than the extent of fibrosis of the lung area conducted within 12 months of first dose.
* Evidence of renal, hepatic, central nervous system, or metabolic dysfunction.
* Evidence of poorly controlled diabetes mellitus (defined as a glycosylated haemoglobin (HbA1c) of > 59 mmol/mol (7.5%).
* Use of systemic immunosuppressants within 30 days of dosing.
* Currently receiving oral steroids, cytotoxic drugs (e.g., chlorambucil, azathioprine, cyclophosphamide, methotrexate), antifibrotic drugs (e.g., pirfenidone), vasodilator therapies for pulmonary hypertension (e.g., bosentan), unapproved (e.g., interferon gamma (INF γ), penicillamine, cyclosporine, mycophenolate) and/or investigational therapies for IPF or administration of such therapies within 4 weeks of initial screening. A current inhaled steroid dose of ≤ 1000 µg beclomethasone dipropionate equivalent per day was acceptable if the dose was anticipated to remain stable during the study.
* History of malignancy, including carcinoma during the preceding 5 years.
* History of, or current asthma.
* Participation in a clinical study of an unlicensed drug in the previous 4 months, or a marketed drug study within the previous 3 months. (N.B. washout period between studies defined as the period of time elapsed between the last dose of the previous study and the first dose of the next study).
* Females of child bearing potential and/or with a positive pregnancy test at the screening visit.

Confirmed at Baseline / Prior to First Dose:

• Development of any exclusion criteria since the screening visit.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2014-09; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Toby Maher, MD, Principal Investigator — Royal Brompton & Harefield NHS Foundation Trust
Locations (5):
- United Kingdom (5):
  - Royal Devon & Exeter Foundation NHS Trust, Exeter, Devon
  - Edinburgh University Hospital, Edinburgh, Scotland
  - The Newcastle Upon Tyne Hospitals NHS Foundation Trust, Newcastle, Tyne and Wear
  - Simbec Research Limited, Merthyr Tydfil, Wales
  - Royal Brompton Hospital, London

IPD SHARING:
Plan to Share IPD: Yes
Interim data from the patient trial will be presented at ICLAF, Dublin 2016

REFERENCES:
- [Derived] Hirani N, MacKinnon AC, Nicol L, Ford P, Schambye H, Pedersen A, Nilsson UJ, Leffler H, Sethi T, Tantawi S, Gravelle L, Slack RJ, Mills R, Karmakar U, Humphries D, Zetterberg F, Keeling L, Paul L, Molyneaux PL, Li F, Funston W, Forrest IA, Simpson AJ, Gibbons MA, Maher TM. Target inhibition of galectin-3 by inhaled TD139 in patients with idiopathic pulmonary fibrosis. Eur Respir J. 2021 May 27;57(5):2002559. doi: 10.1183/13993003.02559-2020. Print 2021 May. PMID 33214209

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 60 subjects were randomised, 39 randomized to treatment, with 24 subjects in Part 1 and 15 subjects in Part 2.
Period: Overall Study
Arm/Group | 0.15 mg TD139 (Part 1) | 1.5 mg TD139 (Part 1) | 3 mg TD139 (Part 1) | 10 mg TD139 Part 1 | 20 mg TD139 Part 1 | 50 mg TD139 Part 1 | Placebo Part 1 | 0.3 mg TD139 Part 2 | 3 mg TD139 Part 2 | 10 mg TD139 Part 2 | Placebo Part 2
Started | 4 | 4 | 4 | 4 | 4 | 4 | 12 | 5 | 5 | 5 | 9
Completed | 4 | 4 | 4 | 4 | 4 | 4 | 12 | 5 | 5 | 4 | 9
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 0.15 mg TD139 (Part 1) | 1.5 mg TD139 (Part 1) | 3 mg TD139 (Part 1) | 10 mg TD139 Part 1 | 20 mg TD139 Part 1 | 50 mg TD139 Part 1 | Placebo Part 1 | 0.3 mg TD139 Part 2 | 3 mg TD139 Part 2 | 10 mg TD139 Part 2 | Placebo Part 2 | Total
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 4 | 12 | 5 | 5 | 5 | 9 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 4 | 4 | 4 | 4 | 4 | 4 | 12 | 1 | 1 | 0 | 0 | 38
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 4 | 5 | 9 | 22
Age, Continuous [Mean (Standard Deviation); unit: Years] | 42.3 (9.07) | 29.8 (6.80) | 39.3 (10.21) | 29.8 (2.06) | 30.8 (9.54) | 32.8 (9.91) | 35.6 (7.53) | 69.0 (6.32) | 73.6 (5.86) | 79.2 (2.77) | 72.9 (4.59) | 50.2 (20.63)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
  Male | 4 | 4 | 4 | 4 | 4 | 4 | 12 | 4 | 5 | 5 | 9 | 59
Region of Enrollment [Number; unit: participants]
  United Kingdom | 4 | 4 | 4 | 4 | 4 | 4 | 12 | 5 | 5 | 5 | 9 | 60

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events
Description: Number of participants reporting Adverse Events from the date of first dose, until 30 days post first dose.
Time Frame: 0 - 30 days
Population: All subjects in Part 1 are included in the safety population. The safety population includes all subjects who received at least one dose of study treatment (TD139 or Placebo). Safety parameters are listed and summarised using descriptive statistics. No formal statistical analysis is planned.
Measure: Count of Participants; unit: Participants
Arm/Group | 0.15 mg TD139 (Part 1) | 1.5 mg TD139 (Part 1) | 3 mg TD139 (Part 1) | 10 mg TD139 Part 1 | 20 mg TD139 Part 1 | 50 mg TD139 Part 1 | Placebo Part 1 | 0.3 mg TD139 Part 2 | 3 mg TD139 Part 2 | 10 mg TD139 Part 2 | Placebo Part 2
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 4 | 12 | 5 | 5 | 5 | 9
Participants | 0 | 0 | 2 | 3 | 4 | 4 | 2 | 4 | 5 | 4 | 7

ADVERSE EVENTS:
Time Frame: Adverse Events are measured from the administration of the first dose, until 30 days post first dose
Arm/Group | 0.15 mg TD139 (Part 1) | 1.5 mg TD139 (Part 1) | 3 mg TD139 (Part 1) | 10 mg TD139 Part 1 | 20 mg TD139 Part 1 | 50 mg TD139 Part 1 | Placebo Part 1 | 0.3 mg TD139 Part 2 | 3 mg TD139 Part 2 | 10 mg TD139 Part 2 | Placebo Part 2
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/4 | 0/4 | 0/4 | 0/4 | 0/4 | 0/12 | 0/5 | 0/5 | 1/5 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/4 | 0/4 | 0/4 | 0/4 | 0/4 | 0/12 | 0/5 | 0/5 | 1/5 | 0/9
Other Adverse Events (participants affected / at risk) | 0/4 | 0/4 | 2/4 | 3/4 | 4/4 | 4/4 | 2/12 | 4/5 | 5/5 | 4/5 | 7/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 0.15 mg TD139 (Part 1) (N=4) | 1.5 mg TD139 (Part 1) (N=4) | 3 mg TD139 (Part 1) (N=4) | 10 mg TD139 Part 1 (N=4) | 20 mg TD139 Part 1 (N=4) | 50 mg TD139 Part 1 (N=4) | Placebo Part 1 (N=12) | 0.3 mg TD139 Part 2 (N=5) | 3 mg TD139 Part 2 (N=5) | 10 mg TD139 Part 2 (N=5) | Placebo Part 2 (N=9)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 0.15 mg TD139 (Part 1) (N=4) | 1.5 mg TD139 (Part 1) (N=4) | 3 mg TD139 (Part 1) (N=4) | 10 mg TD139 Part 1 (N=4) | 20 mg TD139 Part 1 (N=4) | 50 mg TD139 Part 1 (N=4) | Placebo Part 1 (N=12) | 0.3 mg TD139 Part 2 (N=5) | 3 mg TD139 Part 2 (N=5) | 10 mg TD139 Part 2 (N=5) | Placebo Part 2 (N=9)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 4 (4) | 4 (4) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 2 (2)
Abdominal Pain Upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 1 (2)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper Respiratory Tract Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Adrenal Suppression (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (3) | 1 (1)
Vessel Puncture Site Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ear Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Localised Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lower Respiratory Tract Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Flank Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 (0) | 1 (1)
Gout (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal Discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinus Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bladder and Urethral Symptoms (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary Retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper-airway Cough Syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Actinic Keratosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rosacea (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Seborrheic dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Investigators must agree to maintain the confidentiality of the study at all times and must not reveal any information relating to the study without express permission from the study Sponsor.

DOCUMENTS (2):
  • Study Protocol (2016-04-05): https://cdn.clinicaltrials.gov/large-docs/77/NCT02257177/Prot_000.pdf
  • Statistical Analysis Plan (2015-02-05): https://cdn.clinicaltrials.gov/large-docs/77/NCT02257177/SAP_001.pdf